CLINICAL TRIAL: NCT07170501
Title: Postural Control as a Predictor of Disability, Fall-Related Fear, and Social Participation in Elderly Women With Non-Specific Low Back Pain: A Cross-Sectional Study
Brief Title: Postural Control as a Predictor of Disability, Fall-Related Fear, and Social Participation in Elderly Women With Non-Specific Low Back Pain
Status: Completed | Type: Observational
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Azza Mohammed, Assistant professor of Biomechanics, Faculty of Physical Therapy, Cairo University, Cairo University
Other Study IDs: P.T.REC/012/005928; faculty of physical therapy ca (Registry Identifier: faculty of physical therapy)
Record Dates: First submitted 2025-05-19; First posted 2025-09-12 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2025-09

CONDITIONS: Low Back Pain; FALS
Keywords: Postural Control; Disability; Fall-Related fear; Social Participation; Elderly Women ;Non-Specific Low Back Pain
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Non-specific low back pain (NSLBP) is prevalent among elderly women and is often associated with impaired postural control, increased fear of falling, and reduced community participation. Understanding the interplay between these factors is essential for effective rehabilitation and fall prevention strategies in this vulnerable population.

DETAILED DESCRIPTION:
This cross-sectional study aims to investigate

1. the relationship between postural control and its predictive value for fear of falling, disability as measured by the Oswestry Disability Index (ODI), and community integration in elderly women with NSLBP.
2. test whether postural control is a predictor for disability, fall-related fear and social engagement or not.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion criteria include independent ambulation with or without assistive devices and a clinical diagnosis of non-specific low back pain persisting for at least three months.

Exclusion Criteria:

* Participants presenting with specific low back pain due to identifiable organic or pathological causes-such as herniated discs, spinal infections, fractures, tumors, inflammatory arthropathies, or neurological disorders affecting balance or gait-will be excluded to maintain sample homogeneity. Additional exclusion criteria include recent lower limb orthopedic surgery (within the past six months), uncontrolled cardiovascular or metabolic diseases, uncorrected visual or vestibular impairments, and severe cognitive impairment (MMSE < 24).

Ages: 55 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: A total of 70 female participants aged between 55 and 65 years diagnosed with non-specific low back pain will be recruited for this study. All participants will be community-dwelling elderly women with adequate cognitive capacity, confirmed by a Mini-Mental State Examination (MMSE) score of 24 or above, to ensure reliable completion of assessment tools.
Sampling Method: Probability Sample
Enrollment: 70 (Actual)
Dates: Start 2025-05-25 (Actual); Primary Completion 2025-06-30 (Actual); Study Completion 2025-07-03 (Actual)

PRIMARY OUTCOMES:
balance assessed by BBS | three months

SECONDARY OUTCOMES:
disabilty assessed by ODI | three months
Fall-related fear | three months
community integration | three months

CONTACTS AND LOCATIONS:
Locations (1):
- Azza Mohammed, Giza, Egypt

IPD SHARING:
Plan to Share IPD: Undecided
i did not decide